CLINICAL TRIAL: NCT05702008
Title: Social Media as an Information, Education and Communication Tool for Rabies Prevention: An Interventional Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maulana Azad Medical College (Other)
Responsible Party: Principal Investigator, Jay Verma, Principal Investigator, Maulana Azad Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: F.1/IEC/MAMC/90/02/2022/No.112
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Rabies; Health Education; Public Health; Preventive Health Services
MeSH Terms: conditions — Rabies; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The participants in this study arm were administered no intervention.
- Test Group (Experimental): The participants in this arm were administered the following intervention: The test group was administered the rabies IEC material available on the National Center for Disease Control (NCDC) website (https://ncdc.gov.in/index1.php?page=1&ipp=All&lang=1&level=2&sublinkid=502&lid=428) in English and Hindi languages using a WhatsApp broadcast every 3 days for 30 days, in a cyclical manner. This material includes brochures, posters, short films, and informative documents designed to educate the general public about rabies prevention and post-exposure prophylaxis practices. Text messages, encouraging the participants to go through the material, were also a part of this intervention.
  Interventions: Other: Rabies Information Education and Communication Material

INTERVENTIONS:
Other: Rabies Information Education and Communication Material — The test group was administered the rabies IEC material available on the National Center for Disease Control (NCDC) website (https://ncdc.gov.in/index1.php?page=1&ipp=All&lang=1&level=2&sublinkid=502&lid=428) in English and Hindi languages using a WhatsApp broadcast every 3 days for 30 days, in a cyclical manner. This material includes brochures, posters, short films, and informative documents designed to educate the general public about rabies prevention and post-exposure prophylaxis practices. Text messages, encouraging the participants to go through the material, were also a part of this intervention.
  Arms: Test Group

SUMMARY:
Background: Rabies is a fatal disease that can be avoided by treating animal bites promptly. Hence, post-exposure prophylaxis is critical. As a result, the National Rabies Control Program was approved under the 12th five-year plan in India. One of its strategies is to engage in Information, Education and Communication activities. Social media provides an opportunity for the quick and easy dissemination of research but is constrained by a lack of peer review and the risk of misinterpretation. The efficacy of a novel social media-based knowledge dissemination strategy for rabies prevention was tested in this study.

Methods: An experimental study design was followed, wherein 144 preclinical medical students of Maulana Azad Medical College, Delhi, India were included in each control and test group. The test group was administered the intervention, which exposed the participants to health education material via social media across a span of 30 days. Participants' knowledge, attitude and practices were observed before and after the study duration.

ELIGIBILITY:
Inclusion Criteria:

* adult individuals who have a smartphone, internet access and are WhatsApp users
* preclinical medical students, i.e., Bachelor of Medicine, Bachelor of Surgery (MBBS) 1st and 2nd professional year students

Exclusion Criteria:

* individuals who themselves have been a dog bite or rabies victim
* individuals who have a dog bite or rabies victim in the household
* individuals who developed the above criteria during the study duration were excluded from the data analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
To measure the impact of a social media-based dissemination strategy on information dissemination and retention for rabies IEC material among preclinical medical students | 2 months
  The responses obtained through a KAP questionnaire were entered into an MS Excel file and analyzed using SPSS version 24. The responses were scored +1 for the correct answer, -1 for the incorrect answer, and 0 for the "Don't know" answer. Aggregated scores were categorized using Bloom's cut-off points for each of the 3 sections (knowledge, attitude, and practices): "good", if the score was between 80 and 100%, "moderate" if the score was between 60 and 79%, and "poor" if the score was less than 60%. Means and percentages of responses were calculated for both test and control groups, before and after the intervention.
  The changes in responses for both groups were measured and compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Maulana Azad Medical College, Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Breland JY, Quintiliani LM, Schneider KL, May CN, Pagoto S. Social Media as a Tool to Increase the Impact of Public Health Research. Am J Public Health. 2017 Dec;107(12):1890-1891. doi: 10.2105/AJPH.2017.304098. No abstract available. PMID 29116846
- [Result] Aichner T, Grunfelder M, Maurer O, Jegeni D. Twenty-Five Years of Social Media: A Review of Social Media Applications and Definitions from 1994 to 2019. Cyberpsychol Behav Soc Netw. 2021 Apr;24(4):215-222. doi: 10.1089/cyber.2020.0134. Epub 2020 Oct 13. PMID 33847527
- [Result] Cinelli M, Quattrociocchi W, Galeazzi A, Valensise CM, Brugnoli E, Schmidt AL, Zola P, Zollo F, Scala A. The COVID-19 social media infodemic. Sci Rep. 2020 Oct 6;10(1):16598. doi: 10.1038/s41598-020-73510-5. PMID 33024152
- [Result] Dijkstra S, Kok G, Ledford JG, Sandalova E, Stevelink R. Possibilities and Pitfalls of Social Media for Translational Medicine. Front Med (Lausanne). 2018 Dec 6;5:345. doi: 10.3389/fmed.2018.00345. eCollection 2018. PMID 30574495
- [Result] Gatewood J, Monks SL, Singletary CR, Vidrascu E, Moore JB. Social Media in Public Health: Strategies to Distill, Package, and Disseminate Public Health Research. J Public Health Manag Pract. 2020 Sep/Oct;26(5):489-492. doi: 10.1097/PHH.0000000000001096. PMID 32732723
- [Result] Greene JA, Choudhry NK, Kilabuk E, Shrank WH. Online social networking by patients with diabetes: a qualitative evaluation of communication with Facebook. J Gen Intern Med. 2011 Mar;26(3):287-92. doi: 10.1007/s11606-010-1526-3. Epub 2010 Oct 13. PMID 20945113
- [Result] Rajagopalan MS, Khanna VK, Leiter Y, Stott M, Showalter TN, Dicker AP, Lawrence YR. Patient-oriented cancer information on the internet: a comparison of wikipedia and a professionally maintained database. J Oncol Pract. 2011 Sep;7(5):319-23. doi: 10.1200/JOP.2010.000209. Epub 2011 Aug 4. PMID 22211130
- [Result] Eljiz K, Greenfield D, Hogden A, Taylor R, Siddiqui N, Agaliotis M, Milosavljevic M. Improving knowledge translation for increased engagement and impact in healthcare. BMJ Open Qual. 2020 Sep;9(3):e000983. doi: 10.1136/bmjoq-2020-000983. PMID 32943430